CLINICAL TRIAL: NCT01133288
Title: Yulex Glove Prospective Study
Brief Title: Yulex Glove Prospective Study in Spina Bifida
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The funder never paid for the study.
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Charles Curry, Research assistant/co-investigator, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: NA_00024249
Record Dates: First submitted 2010-05-26; First posted 2010-05-28 (Estimated); Results first posted 2011-12-23 (Estimated); Last update posted 2011-12-23 (Estimated); Status verified 2011-11

CONDITIONS: Spina Bifida; Latex Allergy
MeSH Terms: conditions — Spinal Dysraphism; Latex Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Yulex gloves — Study participants will be asked to wear Yulex gloves for routine bowel and bladder care (~30 minutes per day) over a 3 month period.
  Other Names: Yulex Natural Rubber Examination Gloves, Powder-Free; FDA 510(k) Number: K063810

SUMMARY:
This study is to evaluate the safety of Yulex gloves when used by individuals who have documented allergy to natural rubber latex from Hevea brasiliensis. Yulex is a latex from a different plant (Guayule) and in previous studies shows no cross-reactivity to Hevea latex and has not been allergenic in workers exposed to Yulex. The FDA has approved Yulex gloves for use in the general population and has recognized and labeled these gloves as Hevea Latex-free. The labeling still includes a precaution that Yulex gloves may pose a risk for development of allergy because Yulex does contain a small amount of Guayule protein. Yulex Corporation has proposed doing further studies to demonstrate safety and lack of allergenicity in a population that is prone to latex allergy. In the proposed pilot study, the investigators goal is to complete the protocol on 10 adults with spina bifida who are allergic to natural rubber latex who will wear Yulex gloves as part of their regular bladder and bowel care for approximately 30 minutes daily over a 3 month period. The investigators anticipate that the investigators will need to recruit and enroll up to 50 study participants to achieve a final sample of 10 adults with complete study data. Individuals with a history of anaphylaxis will be excluded from the study. The study participants will be tested for Yulex allergy by Glove Puncture Test as well as serology at the beginning and end of the study. The FDA Devices group has reviewed the study design and agreed that this is a suitable first pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with spina bifida between the ages of 18 and 60 who exhibit positive serology to latex (Hevea Brasiliensis).

Exclusion Criteria:

* Possible exclusion criteria include age under 18, does not have spina bifida, or does not exhibit positive serology to latex (Hevea Brasiliensis).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2009-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric B Levey, M.D, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Hugo W. Moser Research Institute at Kennedy Krieger Inc., Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from July 2009 until May 2010. Only 7 participants were enrolled. None of the participants completed the study. Funding was never received from the study sponsor, so the study was terminated.
Pre-assignment Details: Of 7 individuals who enrolled in the study, 2 passed screening and were found to be latex allergic. Funding was never received from the study sponsor and the study was terminated. The 3 month trial of Yulex gloves was not started with any of the participants, so no intervention data is available.
Groups:
- Yulex Glove: Yulex Glove Treatment
Period: Eligibility Assessment
Arm/Group | Yulex Glove
Started | 7
Completed | 2
Not Completed | 5
Not completed — met exclusion criteria | 5
Period: Intervention Allocation
Arm/Group | Yulex Glove
Started | 2
Completed | 0
Not Completed | 2
Not completed — study terminated | 2

BASELINE CHARACTERISTICS:
Arm/Group | Yulex Glove
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 31.3 (6.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Sensitization to Yulex
Description: The primary study outcome will be an assessment for sensitization to Yulex as determined by serological assay for Guayule-specific IgE antibodies. The development of a detectable IgE immune response will be considered a positive study.
Time Frame: Approximately 3 months
Population: No participants were exposed to Yulex because the study was terminated.
Measure: Number; unit: ng/ml
Arm/Group | Yulex Glove
Number analyzed (Participants) | 0

2. Secondary Outcome: Immune Response to Yulex
Description: A secondary study outcome is the development of an immune response to Yulex using a human IgG anti-Guayule immunoassay. The development of a detectable IgG immune response will be considered a positive study.
Time Frame: 3 months
Measure: Number; unit: ug/ml
Arm/Group | Yulex Glove
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were to be assessed over a three month study period. Event data was only assessed on visit one, as none of the participants progressed to visit 2 and no participants received the yulex glove intervention.
Arm/Group | Yulex Glove
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The study was not completed because funding was never received. The two (2/7)enrolled participants who met screening eligibility criteria were terminated early without receiving the yulex glove intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No